CLINICAL TRIAL: NCT06317376
Title: The Effect of Group-based Cardiac Rehabilitation on Pulmonary Function and Aerobic Capacity of Patients With Coronary Artery Bypass Graft Surgery
Brief Title: Group-based Cardiac Rehabilitation on Patients With Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/014131 Maria Haseen
Record Dates: First submitted 2024-01-18; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Post-cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (MICT) (Experimental): MICT 3 session per week with Aerobic exercise on treadmill for 30 minute with moderate intensity.
  Interventions: Other: MICT with Aerobic exercise on treadmill
- control group (standard protocol) (Other): Perform standard hospital protocol 2-3 session per week
  Interventions: Other: standard hospital protocol

INTERVENTIONS:
Other: MICT with Aerobic exercise on treadmill — MICT 3 session per week with Aerobic exercise on treadmill for 30 minute with moderate intensity.
  Arms: experimental group (MICT)
Other: standard hospital protocol — standard hospital protocol
  Arms: control group (standard protocol)

SUMMARY:
1. To determine the effect of Moderate intensity continuous training on Pulmonary function of CABG patients.
2. To determine the effect of MICT on aerobic Capacity of CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females post CABG patients with ages of 40 to 60 years postoperatively.
* The patient with Post Op-Day 5.

Exclusion Criteria:

* Patients who have a history of other Cardiac disorders that interfere with daily life before surgery and those having congenital cardiac anomalies, Tetralogy of Fallot.
* Musculoskeletal and neurological disorders.
* Age more than 60 and less than 40

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Borg rating of perceived exertion scale | 4 weeks
  This scale is used to measure the appearance of the body in the reacttowith the exertion according to the vital sign and symptoms like increased heart rate, respiratory rate, sweating and muscle tiredness. This scale is ranged from 6 to 20 ranking, in thesrankingsng 6 represents "no exertion at all" and twenty reported "maximal exertion during activity". If participants reporta as 12 to 14 score othe n Borg scale this indicate that exertion is at moderate level during exertion. This scale will be used to measure the level of fatigue over all activity of life
6min walk test | 4weeks
  6 min walk test is used to measure the functional status of the individuals. It will be done on both groups to measure the functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Razzaq, MS, Principal Investigator — Riphah International University
Locations (1):
- RMI, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No